CLINICAL TRIAL: NCT06355219
Title: Macrovascular and Microvascular Outcomes in Patients With Type 2 Diabetes and Obesity: Comparison of Metabolic Surgery Versus GLP-1 Receptor Agonists
Brief Title: Macrovascular and Microvascular Morbidity and Mortality After Metabolic Surgery Versus Medicines
Acronym: M6
Status: Completed | Type: Observational
Sponsor: Ali Aminian (Other)
Responsible Party: Sponsor-Investigator, Ali Aminian, Director of the Bariatric and Metabolic Institute, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Other Study IDs: IRB #19-066
Record Dates: First submitted 2024-03-29; First posted 2024-04-09 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes Mellitus; Obesity; Microvascular Disease; Macrovascular Disease; Major Adverse Cardiovascular Events; Nephropathy; Retinopathy; Heart Failure; All Cause Mortality
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Kidney Diseases; Retinal Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metabolic Surgery: Patients aged 18 years to 75 years, who had a BMI ≥30 and T2DM at the time of surgery, and who underwent Roux-en-Y gastric bypass (RYGB) or sleeve gastrectomy (SG) at Cleveland Clinic Health System(CCHS) hospitals in Florida and Ohio between January 1, 2010, and December 31, 2017.
- GLP-1 RAs: Non-surgical patients at CCHS who at randomly assigned index dates had T2DM and obesity, follow-up of at least 30 days after the assigned index date, did not meet any of the exclusion criteria for surgical patients, and did not have metabolic surgery prior to the assigned index date, who continuously received GLP-1 RA for ≥2 years, defined by prescription order for GLP-1 RA placed between January 1, 2010, and December 31, 2017, as well as ≥ 3 documented prescription fills within 1 year before their assigned index date and ≥ 3 fills within 1 year after their index date.

SUMMARY:
The goal of this study is to compare the impact of metabolic surgery and a class of anti-diabetes medications (Glucagon-like peptide-1 receptor agonists,GLP-1 RAs) on occurrence of diseases involving small and large vessels such as heart disease, kidney disease, and disease of the retina (a part of the eye), as well as deaths.

ELIGIBILITY:
Inclusion Criteria:

* BMI>=30 kg/m^2
* Type 2 Diabetes Mellitus
* 18-75 y/o
* Roux-en-Y gastric bypass (RYGB) or sleeve gastrectomy (SG) (Surgical Cohort) at CCHS hospitals in Florida and Ohio between January 1, 2010, and December 31, 2017

For the GLP-1RA Group:

* Follow-up of at least 30 days after the assigned index date
* Did not meet any of the exclusion criteria for surgical patients (see below)
* Did not have metabolic surgery prior to assigned index date.
* Continuously received GLP-1 RA for ≥2 years (prescription order for GLP-1 RA placed between January 1, 2010, and December 31, 2017, as well as ≥ 3 documented prescription fills within 1 year before their assigned index date and ≥ 3 fills within 1 year after their index date)

Exclusion Criteria:

* History of solid organ transplant
* Cardiac ejection fraction <20% any time before index date
* Active cancer
* Cancer code within 1 year before index date
* ED admission within 5 days before index date
* Dialysis or estimated glomerular filtration rate (eGFR) <20 before index date.
* Received care in CCHS locations other than in Ohio and Florida.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with obesity (defined by body mass index [BMI] ≥30 kg/m^2) and T2DM who underwent metabolic surgery at Cleveland Clinic Health System (CCHS) from 2010 to 2017 were compared with similar patients who continuously received GLP-1 RA for at least 2 years. The study used Cleveland Clinic electronic health records (EHR), including Surescripts dispensed prescription records. Follow-up ended on December 31, 2022. To minimize the effects of confounding factors, a doubly robust estimation combining the overlap weighting and outcome regression will be utilized to compare primary and secondary end points in surgical and GLP-1RA groups.
Sampling Method: Probability Sample
Enrollment: 3932 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
All-cause Mortality Rate | After surgical or assigned index date to Dec 31, 2022
  Death from all causes percentage

SECONDARY OUTCOMES:
Incidence of MACE | After surgical or assigned index date to Dec 31, 2022
  Incident major adverse cardiovascular events (MACE, composite of 4 outcomes), defined as the first occurrence of coronary artery events (unstable angina, myocardial infarction, or coronary intervention/surgery), cerebrovascular events (ischemic stroke, hemorrhagic stroke, or carotid intervention/surgery), heart failure, or atrial fibrillation.
Incidence of Nephropathy | After surgical or assigned index date to Dec 31, 2022
  Onset of ≥40% sustained decline in eGFR compared with baseline (calculated using the 2021 CKD-EPI equation), onset of sustained eGFR <15 mL/min/1.73 m^2, initiation of dialysis, or kidney transplant.
Incidence of Retinopathy | After surgical or assigned index date to Dec 31, 2022
  (1) First occurrence of retinopathy in patients who did not have such events at baseline or (2) progression to a more severe form of retinopathy in those with baseline retinopathy

OTHER OUTCOMES:
Incidence of Components of MACE Separately | After surgical or assigned index date to Dec 31, 2022
  Incidence of each of the following MACE components separately: the first occurrence of coronary artery events (unstable angina, myocardial infarction, or coronary intervention/surgery), cerebrovascular events (ischemic stroke, hemorrhagic stroke, or carotid intervention/surgery), heart failure, or atrial fibrillation.
Change in weight percentage | After surgical or assigned index date to Dec 31, 2022
  Relative change in weight percentage at follow up compared to index date
Change HBA1c percentage | After surgical or assigned index date to Dec 31, 2022
  Absolute change HBA1c percentage at follow up compared to index date
Trends of prescription and dispenses of medications for T2DM and cardio-vascular conditions | After surgical or assigned index date to Dec 31, 2022
  Using dates of prescription orders and dispenses of medications for T2DM and cardio-vascular conditions
Progression of Chronic Kidney Disease (CKD) in Patients with CKD stages 3 and 4 at baseline | After surgical or assigned index date to Dec 31, 2022
  Defined as onset of ≥ 50% sustained decline in eGFR compared with baseline, onset of sustained eGFR <15 mL/min/1.73 m2, initiation of dialysis, or kidney transplant after the index date.
Cost-effectiveness of Metabolic Surgery vs GLP-1RAs | After surgical or assigned index date to Dec 31, 2022
  Defined as the cost per life year and the cost per quality adjusted life year (QALY) in the surgical and nonsurgical patients.
Incidence of Adverse Events After Metabolic Surgery | 90 days after surgical index date
  Serious complications following surgery include bleeding requiring transfusion, pulmonary adverse events, venous thromboembolism, cardiac events, renal failure requiring dialysis, gastrointestinal leak, bowel obstruction requiring surgery, gastric/anastomotic stricture or ulcer, and sepsis.

IPD SHARING:
Plan to Share IPD: No